CLINICAL TRIAL: NCT04383379
Title: Evidence-Based Practice for Improving Quality(EPIQ) to Improve the Rate of Mother's Own Milk Feeding of Premature Infants in NICU: Study Protocol for a Cluster Randomized Controlled Trial
Brief Title: To Improve the Rate of Mother's Own Milk Feeding of Premature Infants in NICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Collaborators: Nanjing Maternity and Child Health Care Hospital (Other); Jiangsu Maternity and Child Health Care Hospital (Unknown); Xuzhou Maternity and Child Health Care Hospital (Other); Affiliated Hospital of Jiangsu University (Other); Yangzhou Maternity and Child Health Care Hospital (Unknown); Lianyungang Maternity and Child Health Care Hospital (Unknown); Nantong Maternity and Child Health Care Hospital (Unknown); The First People's Hospital of Jiangyin (Unknown); Yangzhou No.1 People's Hospital (Other); Subei people's Hospital (Unknown); Wuxi Maternity and Child Health Care Hospital (Unknown); The Affiliated Hospital of Xuzhou Medical University (Other); Changzhou Maternal and Child Care Hospital (Other)
Responsible Party: Principal Investigator, Zhangbin Yu, Principal Investigator of Nan Jing Maternity and Child Health Care Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NMU-FY2016-73
Record Dates: First submitted 2020-05-07; First posted 2020-05-12 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Quality Improvement; Breast-feeding; Premature Infant
Keywords: Quality Improvement; breast-feeding; premature infant; cluster randomized controlled
MeSH Terms: conditions — Breast Feeding; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 6 NICUs in the intervention group . The participating units of the intervention group determine the improvement items (one or more) in each quarter from the list of best practices of breast feeding quality improvement of Jiangsu Province, and report the improvement plan to the supervision unit, and recommend the application of PDSA (plan-do-study-act) for the implementation of quality improvement loop. Report the implementation of quality improvement to the supervision unit on a quarterly basis.
  Interventions: Behavioral: Experimental: Intervention group
- control group (No Intervention): Continue current practices

INTERVENTIONS:
Behavioral: Experimental: Intervention group — The intervention NICUs (n = 6) will receive training in the Evidence-based Practice for Improving Quality (EPIQ) method and then develop, implement, and document evidence-based practice changes toimprove the rate of breastfeeding . Compliance with practice changes and neonatal outcomes will be monitored. NICUs will receive quarterly feedback on their progress, as well as access to implementation support.
  Arms: Intervention group

SUMMARY:
Thirteen hospitals in China will participate in the study, which objectives of this study is to improve the rate of mother's own milk feeding of premature infants in neonatal intensive care unit(NICU), evaluate the effectiveness of improving the quality of breastfeeding in clinical use ,form standardized process and improve clinical medical quality of premature infants.

DETAILED DESCRIPTION:
In this study, the cluster randomized controlled matching design was used. Considering that evidence-based practice for improving quality(EPIQ) method is not only to improve the quality of individual, but also to improve the quality of breast-feeding of the whole neonatal intensive care unit(NICU), so a hospital was chosen as a cluster. The supervision unit is used for the quality control , coordination and technical support in the whole study process.The two NICU with similar number of premature infants, the same scale of NICU and little difference in the recognition of breast-feeding quality improvement measures that meet the inclusion criteria are taken as the a floor, and then randomly divided into two groups, taking the NICU as intervention group or the control group can avoid the individual influence of the intervention. In this study, recruited 12 NICUs. The purpose of study is to to increase the consumption of mother's own milk of premature infants through the existing measures of improving the breastfeeding quality, and then to improve the quality of life of the premature infant, and to further evaluate whether this model of improving the breastfeeding quality can be promoted in other NICU.

ELIGIBILITY:
Inclusion Criteria:

* Weight less than 1500g or gestational age less than 32 weeks;
* Admission to NICU.

Exclusion Criteria:

* Pregnancy with serious diseases, infectious diseases or other medical contraindications for breast-feeding (such as galactosemia);
* infants did not survive were excluded.

Max Age: 120 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1500 (Estimated)
Dates: Start 2020-05-15 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
exclusive breastfeeding rate 24 hours before discharge | two years
  exclusive breastfeeding rate 24 hours before discharge

SECONDARY OUTCOMES:
Time of Mother's Own Milk at starting feed（hours） | two years
  Time of Mother's Own Milk at starting feed（hours）
Proportion of first time Mother's Own Milk (%) | two years
  Proportion of first time Mother's Own Milk (%)
Duration of parenteral nutrition (days) | two years
  Duration of parenteral nutrition (days)
Time to total gastrointestinal feeding (days) | two years
  Time to total gastrointestinal feeding (days)
Pump milk times (times /d) and amount (ml / d) ：1-3d, 4-7d ,8-14d | two years
  Pump milk times (times /d) and amount (ml / d) ：1-3d, 4-7d ,8-14d

CONTACTS AND LOCATIONS:
Overall Officials: Han Shuping, PhD, Study Director — Nanjing Maternity and Child Health Care Hospital; Yu Zhangbin, PhD, Study Director — Nanjing Maternity and Child Health Care Hospital; Chen Xiaoqing, PhD, Principal Investigator — Jiangsu Maternity and Child Health Care Hospital; Deng Xiaoyi, PhD, Principal Investigator — Xuzhou Maternity and Child Health Care Hospital; Lu Hongyan, PhD, Principal Investigator — Affiliated Hospital of Jiangsu University; Wu Xinping, PhD, Principal Investigator — Yangzhou Maternity and Child Health Care Hospital; Gao Yan, PhD, Principal Investigator — Lianyungang Maternity and Child Health Care Hospital; Li Shuangshuang, PhD, Principal Investigator — Nantong Maternity and Child Health Care Hospital; Wan Jun, PhD, Principal Investigator — The First People's Hospital of Jiangyin; Wu Mingfu, PhD, Principal Investigator — Yangzhou No.1 People's Hospital; Zhu Lingling, PhD, Principal Investigator — Subei people's Hospital; Zhou Qin, PhD, Principal Investigator — Wuxi Maternity and Child Health Care Hospital; Wang Jun, PhD, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University; Wang Huaiyan, PhD, Principal Investigator — Changzhou Maternal and Child Care Hospital
Locations (1):
- Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Huo J, Wu X, Gu C, Yu Z, Zhang J, Chen X, Zhu J, Liu F, Liu B, Li Q, Han S. Using a WeChat mini-program-based lactation consultant intervention to increase the consumption of mother's own milk by preterm infants in the neonatal intensive care unit: a study protocol for a cluster randomized controlled trial. Trials. 2021 Nov 24;22(1):834. doi: 10.1186/s13063-021-05731-6. PMID 34819117